CLINICAL TRIAL: NCT06328894
Title: A Randomized Controlled Trial to Explore the Effect of Different Feeding Modes on Psychological Condition and Experience in Stroke Patients
Brief Title: Effect of Different Feeding Modes on Psychological Condition and Experience in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IOE Psychological
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comprehensive rehabilitation therapy+Intermittent Oro-esophageal Tube Feeding (Experimental): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  The observation group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- comprehensive rehabilitation therapy+Nasogastric Tube Feeding (Active Comparator): Assigned randomly before the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Besides, the control group was given enteral nutritional support with Nasogastric Tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Nasogastric Tube Feeding — Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Arms: comprehensive rehabilitation therapy+Nasogastric Tube Feeding
Device: Intermittent Oro-esophageal Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: comprehensive rehabilitation therapy+Intermittent Oro-esophageal Tube Feeding
Behavioral: comprehensive rehabilitation therapy — Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Pulmonary function training, including standing training, cough training, and diaphragm muscle training.

SUMMARY:
The goal of this clinical trial is to compare the differences on Psychological Condition and Experience in ischemic stroke patients using Intermittent Oro-esophageal Tube and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare Psychological Condition and Experience of two groups.

DETAILED DESCRIPTION:
The study will last 15 days for each participant. The goal of this clinical trial is to compare the differences on Psychological Condition and Experience in ischemic stroke patients using Intermittent Oro-esophageal Tube and Nasogastric Tube. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the control group will use Nasogastric Tube. Researchers will compare Psychological Condition and Experience of two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | day 1 and day 15 and day 60
  The Hospital Anxiety and Depression Scale was used to assess the participants' anxiety and depression symptoms. The scale includes two subscales: anxiety and depression, each consisting of 7 items. Each item is scored from 0 to 3. The total score for each subscale could range between 0 and 21. A higher total score indicates more severe symptoms.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Adult Profile | day 1 and day 15 and day 60
  The Patient-Reported Outcomes Measurement Information System Adult Profile was used to assess subjective social isolation This assessment includes 8 items, each scored between 1 and 5. The total score could range from 8 to 40, with higher scores indicating worse subjective social isolation.
Stroke Self-Efficacy Questionnaire | day 1 and day 15 and day 60
  The Stroke Self-Efficacy Questionnaire was used to assess self-efficacy in functional independence and self-management.The Stroke Self-Efficacy Questionnaire includes 13 items, each scored between 0 and 10. The total score could range from 0 to 130. A higher score indicates better self-efficacy.
Visual Analog Scale for Fatigue | day 1 and day 15 and day 60
  The Visual Analog Scale for Fatigue is used to assess fatigue. It is a horizontal line from 0 to 4. The total score could range from 0 to 4, with higher scores indicating more fatigue.
Visual Analog Scale for Nausea | day 1 and day 15 and day 60
  The Visual Analog Scale for Nausea was used to assess recent perceived nausea. It is a horizontal line from 0 to 10, where 0 indicates no nausea and 10 represents unbearable nausea, with higher scores indicating more unbearable nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Study Chair — Site Coordinator of United Medical Group
Locations (2):
- China (2):
  - Department of rehabilitation medicine, the first ZU hospital north campus, Zhenzhou
  - Department of rehabilitation medicine, the first ZU hospital western campus, Zhenzhou